CLINICAL TRIAL: NCT02552082
Title: The Verification Study on the Effectiveness of Rotational Tolerance of Scorpio NRG Study in TKA
Brief Title: Scorpio Non Restricted Geometry (NRG) Study in Japan
Status: Completed | Type: Observational
Sponsor: Stryker Japan K.K. (Industry)
Responsible Party: Sponsor
Other Study IDs: SJCR-OR-1501
Record Dates: First submitted 2015-08-10; First posted 2015-09-16 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Scorpio NRG
  Interventions: Device: Scorpio NRG posterior stabilized (PS)

INTERVENTIONS:
Device: Scorpio NRG posterior stabilized (PS)

SUMMARY:
The purpose of this study is to evaluate the range of motion (ROM), mid-flexion stability (gap balance), and implant position (size and angle) for the Scorpio NRG device. Relationship between these parameters and clinical outcomes will be evaluated as well as the importance of rotational tolerance. It is expected that the Scorpio NRG will have good clinical outcomes and perform the same or better than other total knee implants.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is candidate for primary total knee arthroplasty (TKA).
2. Patient who has diagnosis of osteoarthritis or rheumatoid arthritis.
3. Patient who is age 20 or over.
4. Patient who signed an Institutional Review Board (IRB)-approved, study specific Informed Patient Consent Form.
5. Patient who is willing and able to comply with postoperative scheduled evaluations.

Exclusion Criteria:

1. Patient who has a bacterial infectious disease or has a risk high of a bacterial infection.
2. Patient who requires revision surgery.
3. Patient who is morbidly obese, defined as having a Body Mass Index (BMI) > 40.
4. Patient who is or may be pregnant female.
5. Patient who has a neuromuscular or neurosensory deficiency, which limits ability to evaluate the safety and efficacy of the device.
6. Patient with diagnosed systemic disease (i.e. Paget's disease, renal osteodystrophy).
7. Patient who is immunologically suppressed or receiving chronic steroids.
8. Patient who is judged ineligible with specific reason by primary doctor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who has diagnosis of osteoarthritis or rheumatoid arthritis.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in Range of motion(ROM) | Pre-operation, intraoperative, 6 months and 1 year after surgery

SECONDARY OUTCOMES:
Change in Japanese Orthopaedics Association (JOA) score, | Pre-operation, intraoperative, 6 months and 1 year after surgery
Change in Knee Society Score (KSS) | Pre-operation, intraoperative, 6 months and 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fukuoka Tokushukai Hospital., Kasuga, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No